CLINICAL TRIAL: NCT03164603
Title: A Phase 1 Study of NLG802 for Adult Patients With Recurrent Advanced Solid Tumors
Brief Title: NLG802 Indoleamine 2,3-Dioxygenase (IDO) Inhibitor in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLG8021
Record Dates: First submitted 2017-05-22; First posted 2017-05-23 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NLG8021 Dose Escalation (Experimental): Approximately 6 to 36 participants will be enrolled and treated at escalating doses of NLG802. Treatment may continue until unacceptable toxicity or disease progression. Successive groups of at least 3 participants will be evaluated during a 28-day window for DLTs, which will determine the enrollment and dosing for subsequent cohorts in the dose-escalation stage.
  Interventions: Drug: NLG802

INTERVENTIONS:
Drug: NLG802 — Indoleamine 2,3-Dioxygenase (IDO) Inhibitor

SUMMARY:
This is an open-label Phase I study to evaluate the safety, tolerability, and pharmacokinetics of escalating oral doses of NLG802, an investigational agent intended to inhibit the indoleamine 2,3-dioxygenase 1 (IDO1) enzyme and help the human immune system attack solid tumor cells more effectively.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed solid tumor cancer (including glioblastoma)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic and organ function

Exclusion Criteria:

* Active or history of medically significant autoimmune disease
* Cytotoxic therapy or investigational agent use within 28 days
* Human immunodeficiency virus (HIV), active hepatitis B or C
* Untreated brain metastases
* Known QT interval prolongation
* Use of concomitant medications with high risk of causing Torsades des Pointes.
* Use of immune suppressive agents within 30 days
* More than one active malignancy at the time of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-06-29 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with dose-limiting toxicities | 28 Days
Percentage of patients with adverse events | From Screening until 30 days after last dose (up to approximately 2 years)

SECONDARY OUTCOMES:
Pharmacokinetics: Serum concentrations (Cmax/Steady State) | 21 Days
Percentage of Participants With Objective Response According to Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) as Determined by the Investigator | From Screening until disease progression, death, new anti-cancer therapy, or premature study withdrawal (up to approximately 3 years)
Percentage of Participants With Progression Free Survival (PFS) | 18 months
  equals date of progression/death - date of study enrollment

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Florida, Gainesville, Florida
  - Washington University School of Medicine, St Louis, Missouri
  - University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico

IPD SHARING:
Plan to Share IPD: No